CLINICAL TRIAL: NCT00888264
Title: A 6 Month Observational Multicentric Prospective Study Observing the Use of Atypical Antipsychotics in Patients Diagnosed With Bipolar I or II Disorder, in the Course of a Major Depressive Episode
Brief Title: A NIS Evaluating the Treatment Patterns of Atypical Antipsychotics in Patients Diagnosed With Bipolar I or II Disorder
Acronym: HARMONY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MCMD, AstraZeneca
Other Study IDs: NIS-NBE-SER-2008/1
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Bipolar Disorders
Keywords: Antipsychotics; Bipolar Disorder; Depressive episodes; Bipolar I or II Disorders
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this NIS is to obtain data on how AAPs are used in DSM-IV-TR Bipolar I and II Disorder, in the course of a major depressive episode. Both the parameters of use of AAPs and clinical evaluation will be recorded and potential differences that may exist due to epidemiological factors or comorbidities will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, diagnosed with Bipolar I or II Disorder, having presented or presenting a major depressive episode (according to DSM-IV-TR) with a starting date of 6 months maximum before the inclusion.
* Current treatment with atypical antipsychotic(s) (AAP(s)) minimal 1 month and maximum 6 months prior to the first study visit
* Patient takes an AAP at an adequate therapeutic dose as indicated in the local Summary of Product Characteristics (SPC) and current medical practice

Exclusion Criteria:

* Patients diagnosed with Bipolar I or II, experiencing a hypomanic, manic or mixed episode at time of inclusion
* Pregnant or breastfeeding women, or women of childbearing potential not using a medical reliable method of contraception as stated in the SPC of the AAPs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients (male or female), diagnosed with Bipolar I or II disorder, having presented or presenting a major depressive episode (according to DSM-IV-TR) with starting date of 6 months maximum before the inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Details of any AAP prescribed 1 to 6 months prior to the first study visit: | 4 visits

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS), a 10-point observer rating scale, used to assess the symptoms and severity of depression. | 4 visits
Young Mania Rating Scale (YMRS), an 11-point observer rating scale, used to assess the symptoms and severity of mania. | 4 visits
Remission rate for the major depressive episode, in progress at inclusion | At completion

CONTACTS AND LOCATIONS:
Locations (45):
- Belgium (45):
  - Research Site, Aarschot
  - Research Site, Afsnee
  - Research Site, Antwerp
  - Research Site, Asse
  - Research Site, Berchem
  - Research Site, Bertrix
  - Research Site, Bierbeek
  - Research Site, Bouge
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Dave
  - Research Site, Dendermonde
  - Research Site, Erpe Mere
  - Research Site, Geel
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Ixelles-Elsene
  - Research Site, Kortenberg
  - Research Site, Kortrijk
  - Research Site, Laken
  - Research Site, Lebbeke
  - Research Site, Lede
  - Research Site, Leuven
  - Research Site, Libramont
  - Research Site, Lierneux
  - Research Site, Liège
  - Research Site, Lubbeek
  - Research Site, Malle
  - Research Site, Marchienne-au-Pont
  - Research Site, Mons
  - Research Site, Montignies-sur-Sambre
  - Research Site, Namur
  - Research Site, Ottignies
  - Research Site, Roselaere
  - Research Site, Saint Denijs Westrem
  - Research Site, Saint-Servais
  - Research Site, Sint-Josse-ten-Noode
  - Research Site, Sint-Martens-Latem
  - Research Site, Sint-Niklaas
  - Research Site, Sleidinge
  - Research Site, St-Truiden
  - Research Site, Tienen
  - Research Site, Tournai
  - Research Site, Zottegem
  - Research Site, Zoutleeuw